CLINICAL TRIAL: NCT06018337
Title: A Phase 3, Randomized, Multi-center, Open-Label Study of DB-1303 Versus Investigator's Choice Chemotherapy in Human Epidermal Growth Factor Receptor 2 (HER2)-Low, Hormone Receptor Positive (HR+) Metastatic Breast Cancer Patients Whose Disease Has Progressed on Endocrine Therapy (ET) (DYNASTY-Breast02)
Brief Title: A Study of DB-1303/BNT323 vs Investigator's Choice Chemotherapy in HER2-Low, Hormone Receptor Positive Metastatic Breast Cancer (DYNASTY-Breast02)
Status: Recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: DualityBio Inc. (Industry)
Collaborators: BioNTech SE (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: DB-1303-O-3002; CTR20233708 (Other: CENTER FOR DRUG EVALUATION, NMPA)
Record Dates: First submitted 2023-08-25; First posted 2023-08-30 (Actual); Last update posted 2025-07-18 (Actual); Status verified 2025-02

CONDITIONS: Metastatic Breast Cancer
Keywords: HER2-low; IHC 2+; BC; Breast Cancer
MeSH Terms: conditions — Breast Neoplasms | interventions — Capecitabine; Paclitaxel; 130-nm albumin-bound paclitaxel

STUDY DESIGN:
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- DB-1303/BNT323 (Experimental): Enrolled Subjects will be randomized to receive a 8 mg/kg IV dose of DB-1303/BNT323 on Day 1 of each cycle Q3W
  Interventions: Drug: DB-1303/BNT323
- investigator's choice single agent chemotherapy (Active Comparator): Enrolled Subjects will be randomized to receive investigator's choice single agent chemotherapy (capecitabine:1000 or 1250 mg/m2, Oral, Twice daily orally for 2 weeks followed by a 1-week rest period in 3-week cycles; paclitaxel：80 mg/m2， IV, Every week (QW) in 3-week cycles; or nab-paclitaxel: 100 mg/m2, IV, Every week (QW) for 3 weeks followed by a one-week rest period in 4-week cycles) until RECIST 1.1 defined disease progression (PD), unless there is unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met.
  Interventions: Drug: Capecitabine; Drug: Paclitaxel; Drug: Nab-paclitaxel

INTERVENTIONS:
Drug: DB-1303/BNT323 — IV
  Arms: DB-1303/BNT323
Drug: Capecitabine — Oral
  Arms: investigator's choice single agent chemotherapy
Drug: Paclitaxel — IV
  Arms: investigator's choice single agent chemotherapy
Drug: Nab-paclitaxel — IV
  Arms: investigator's choice single agent chemotherapy

SUMMARY:
The goal of this clinical trial is to assess the efficacy of DB-1303/BNT323 compared with investigator's choice chemotherapy in terms of progression-free survival (PFS) by blinded independent central review (BICR) in the HR+, HER2-low (immunohistochemistry [IHC]2+/in situ hybridization [ISH]- and IHC 1+) population.

DETAILED DESCRIPTION:
The study is a Phase III, Randomized, Multi-center, Open-label study in HER2-low, HR+ metastatic breast cancer subjects whose disease has progressed on at least 2 lines of prior ET or within 6 months of first line ET + Cyclin-dependent kinase (CDK) 4/6 inhibitor in the metastatic setting. The primary purpose of the study is to determine the efficacy and safety of DB-1303/BNT323 compared with investigator's choice single agent chemotherapy in the target population. Approximately 532 subjects with HER2 IHC 2+/ISH- and IHC 1+ (HER2-low] expression will be randomized 1:1 across approximately 255 centers globally to receive either DB-1303 or investigator's choice single agent chemotherapy (capecitabine, paclitaxel or nab-paclitaxel) until Response Evaluation Criteria in Solid Tumors (RECIST) 1.1 defined disease progression (PD), unless there is unacceptable toxicity, withdrawal of consent, or another criterion for discontinuation is met.

ELIGIBILITY:
Inclusion Criteria:

1. Male or female adults (defined as ≥ 18 years of age or acceptable age according to local regulations at the time of voluntarily signing of informed consent).

2. Pathologically documented breast cancer that:

1. Is advanced or metastatic
2. Has HER2-low expression (IHC 1+ or IHC 2+/ISH-) as determined by the central laboratory result.
3. Was never previously reported as HER2-positive (IHC 3+ or ISH+) as per American Society of Clinical Oncology/College of American Pathologists (ASCO/CAP) guidelines.
4. Is documented as HR+ (either estrogen receptor [ER] and/or progesterone receptor [PgR] positive [ER or PgR ≥1%]) per ASCO/CAP guidelines (Allison et al 2020).

3. Must have an adequate tumor tissue sample available for assessment of HER2 by central laboratory, in formalin fixation and paraffin embedding (FFPE) blocks based on a mandatory FFPE tumor sample preferably obtained at the time of metastatic disease or later;

4. Eastern Cooperative Oncology Group performance status of 0 or 1.

5. Must have had either:

1. Disease progression on endocrine therapy + CDK4/6 inhibitor within 6 months of starting first line treatment for metastatic disease and considered appropriate for chemotherapy as the next treatment by the investigator, OR
2. Disease progression on at least 2 previous lines of ET with or without a targeted therapy (such as CDK4/6, mammalian target of rapamycin [mTOR] or phosphoinositide 3-kinase [PI3-K] inhibitors) administered for the treatment of metastatic disease.

6. No prior chemotherapy for advanced or metastatic breast cancer. Subjects who have received chemotherapy in the neo-adjuvant or adjuvant setting are eligible, as long as they have had a disease-free interval (defined as completion of systemic chemotherapy to diagnosis of advanced or metastatic disease) of >12 months.

7. Life expectancy ≥12 weeks at screening.

8. Subjects must have at least one measurable lesion as defined per RECIST v1.1 (For bone only disease, subjects with lytic or mixed lytic bone lesions that can be measured by CT or MRI are eligible; subjects with sclerotic/osteoblastic bone lesions are not eligible).

9. Has LVEF ≥ 50% by either echocardiography (ECHO) or multiple-gated acquisition (MUGA) within 28 days before randomization.

10. Adequate organ and bone marrow function within 14 days before randomization.

11. Has adequate treatment washout period before randomization.

12. Evidence of post-menopausal status or negative serum pregnancy test for females of childbearing potential who are sexually active with a non-sterilized male partner. For women of childbearing potential, a negative result for serum pregnancy test (test must have a sensitivity of at least 25 mIU/mL) must be available at the screening visit and urine beta-human chorionic gonadotropin (β-HCG) pregnancy test prior to each administration of study treatment.

Women of childbearing potential are defined as those who are not surgically sterile (i.e., underwent bilateral salpingectomy, bilateral oophorectomy, or complete hysterectomy) or post-menopausal.

13. Female subjects of childbearing potential who are sexually active with a non-sterilized male partner must use at least one highly effective method of contraception from the time of screening and must agree to continue using such precautions for 7 months after the last dose of study treatment. Not all methods of contraception are highly effective. Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the subject for the duration of the study treatment and the drug washout period (7 months). Periodic abstinence (e.g., calendar ovulation, symptothermal, post ovulation methods), the rhythm method, and the withdrawal method are not acceptable methods of contraception. Female subjects must not donate ova, or retrieve for their own use, from the time of screening and throughout the study treatment period, and for at least 7 months after the last dose of study treatment. They should refrain from breastfeeding throughout this time. Preservation of ova may be considered prior to randomization in this study.

14. Non-sterilized male subjects who are sexually active with a female partner of childbearing potential must use a condom with spermicide from screening and throughout the duration of the study treatment and the washout period (4 months after the last dose of DB-1303, 6 months after the last dose of paclitaxel or nab-paclitaxel, and 3 months after the last dose of capecitabine). Abstinence is acceptable only as true abstinence when this is in line with the preferred and usual lifestyle of the subject for the duration of the study treatment and the drug washout period. Periodic abstinence (e.g., calendar ovulation, symptothermal, post ovulation methods), the rhythm method, and the withdrawal method are not acceptable methods of contraception. It is strongly recommended for the female partners of a male subject also use at least one highly effective method of contraception throughout this period. In addition, male subjects should refrain from fathering a child or donating sperm throughout the duration of the study and the washout period (4 months after the last dose of DB-1303, 6 months after the last dose of paclitaxel or nab paclitaxel, and 3 months after the last dose of capecitabine). Preservation of sperm should be considered prior to randomization in this study.

15. Must be able and willing to comply with the protocol requirements and must sign and date the informed consent form prior to any screening evaluations.

Exclusion Criteria:

1. Ineligible for all options in the investigator's choice chemotherapy arm.
2. Uncontrolled intercurrent illness, including but not limited to, ongoing or active infection, uncontrolled or significant cardiovascular disease, serious chronic gastrointestinal conditions associated with diarrhea, or psychiatric illness/social situations that would limit compliance with study requirement, substantially increase risk of incurring adverse events or compromise the ability of the subject to give written informed consent.
3. Clinically uncontrolled pleural effusion, ascites or pericardial effusion requiring repeated drainage, peritoneal shunt or cell-free concentrated ascites reinfusion therapy within 2 weeks prior to the randomization.
4. Uncontrolled or significant cardiovascular disease
5. Has a medical history of interstitial lung diseases (e.g., non-infectious interstitial pneumonia, pneumonitis, pulmonary fibrosis, and radiation pneumonitis which needs glucocorticoids and antibiotics) or current interstitial lung diseases or who are suspected to have these diseases by imaging at screening.
6. Has unresolved toxicities from previous anticancer therapy, defined as toxicities (other than alopecia) not yet resolved to Grade ≤ 1 or baseline or Grade ≤ 2 anemia.
7. Previous treatment with anti-HER2 therapy.
8. Prior treatment with antibody-drug conjugate that comprised an exatecan derivative that is a topoisomerase I inhibitor.
9. Prior randomization or treatment in a previous DB-1303/BNT323 study regardless of treatment assignment.
10. Has substance abuse or any other medical conditions such as psychological conditions, that may, in the opinion of the Investigator, interfere with the subject's participation in the clinical study or evaluation of the clinical study results.
11. Individuals who are dependent on the Sponsor, clinical site, or Investigator (e.g., is an employee of the Sponsor or the clinical trial site, a dependent of the Investigator, or any site staff member otherwise supervised by the Investigator).
12. Individuals who are committed to an institution by virtue of an order issued either by the judicial or the administrative authorities, in accordance with local regulations.

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 532 (Estimated)
Dates: Start 2024-01-18 (Actual); Primary Completion 2026-05 (Estimated); Study Completion 2028-07 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival (PFS) in the HR+, HER2-low population | Up to approximately 51 months
  PFS by BICR according to RECIST 1.1 in the HR+, HER2-low population

SECONDARY OUTCOMES:
Overall survival (OS) in the HR+, HER2-low population | Up to approximately 51 months
  OS in the HR+, HER2-low population
Objective response rate (ORR) in the HR+, HER2-low population | Up to approximately 51 months
  ORR by BICR and Investigator assessment according to RECIST 1.1 in the HR+, HER2-low population
PFS by Investigator assessment | Up to approximately 51 months
  PFS by Investigator assessment according to RECIST 1.1 in the HR+, HER2-low population
Duration of response (DoR) in the HR+, HER2-low population | Up to approximately 51 months
  DoR by BICR and Investigator assessment according to RECIST 1.1 in the HR+, HER2-low population
Treatment-emergent adverse events (TEAEs) | from the time of the subject signing the informed consent form (ICF) until the follow-up period is completed (35 days after the last dose of study treatment
  TEAEs per National Cancer Institute (NCI) Common Terminology Criteria for Adverse Events (CTCAE) v5.0
Serious adverse events (SAEs) | from the time of the subject signing the ICF until the follow-up period is completed (35 days after the last dose of study treatment
  SAEs per NCI CTCAE v5.0
Patient reported outcomes (PROs): European Organization for Research and Treatment of Cancer (EORTC) Quality of Life Questionnaire (QLQ) - C30 | Up to approximately 51 months
  Change from baseline in the functioning/symptom/global quality of life (QoL) subscales of EORTC QLQ-C30. Scale scores range from 0-100. For functioning and global QoL scales, higher scores indicate better functioning or global health status. For symptom scales, higher scores indicate greater symptom burden.
Patient reported outcomes (PROs): EORTC QLQ-BR45 | Up to approximately 51 months
  Change from baseline in the functioning/symptom subscales of EORTC QLQ-BR45. Scale scores range from 0-100. For functioning scales, higher scores indicate better functioning. For symptom scales, higher scores indicate greater symptom burden.
Patient reported outcomes (PROs): European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) | Up to approximately 51 months
  Change from baseline in EQ-5D-5L health state utility index score and Visual Analogue Scale (VAS) score. VAS score range from 0-100, higher scores indicate better health status.
European Quality of Life Five Dimension Five Level Scale (EQ-5D-5L) | Up to approximately 51 months
  EQ-5D-5L health state utility index score and Visual Analogue Scale (VAS) score. The change from baseline value will be reported.

CONTACTS AND LOCATIONS:
Overall Officials: Joyce O'Shaughnessy, PHD, Principal Investigator — Texas Oncology - Baylor Charles A. Sammons Cancer center
Locations (253):
- United States (42):
  - Research Site 1141-0, Tucson, Arizona
  - Research Site 1114-0, Fullerton, California
  - Research Site 1107-0, Los Angeles, California
  - Research Site 1118-0, Orange, California
  - Research Site 1143-0, Sacramento, California
  - Research Site 1132-0, Santa Barbara, California
  - Research Site 1137-0, Aurora, Colorado
  - Research Site 1129-0, Lone Tree, Colorado
  - Research Site 1154-0, Jacksonville, Florida
  - Research Site 1145-0, Miami, Florida
  - Research Site 1150-0, Orange City, Florida
  - Research Site 1125-0, Palm Bay, Florida
  - Research Site 1110-0, Savannah, Georgia
  - Research Site 1147-0, Chicago, Illinois
  - Research Site 1124-0, Chicago Ridge, Illinois
  - Research Site 1152-0, Fort Wayne, Indiana
  - Research Site 1106-0, Merriam, Kansas
  - Research Site 1104-0, Louisville, Kentucky
  - Research Site 1122-0, Silver Spring, Maryland
  - Research Site 8639-0, Silver Spring, Maryland
  - Research Site 1109-0, Kansas City, Missouri
  - Research Site 1111-0, Florham Park, New Jersey
  - Research Site 1157-0, Santa Fe, New Mexico
  - Research Site 1148-0, Staten Island, New York
  - Research Site 1105-0, Westbury, New York
  - Research Site 1144-0, Chapel Hill, North Carolina
  - Research Site 1138-0, Akron, Ohio
  - Research Site 1160-0, Cincinnati, Ohio
  - Research Site 1133-0, Eugene, Oregon
  - Research Site 1126-0, Tigard, Oregon
  - Research Site 1134-0, Broomall, Pennsylvania
  - Research Site 1123-0, Horsham, Pennsylvania
  - Research Site 1149-0, Knoxville, Tennessee
  - Research Site 1102-0, Nashville, Tennessee
  - Research Site 1101-0, Dallas, Texas
  - Research Site 1116-0, Denison, Texas
  - Research Site 1115-0, Houston, Texas
  - Research Site 1117-0, San Antonio, Texas
  - Research Site 1130-0, Salt Lake City, Utah
  - Research Site 1108-0, Fairfax, Virginia
  - Research Site 1131-0, Fairfax, Virginia
  - Research Site 1127-0, Roanoke, Virginia
- Argentina (12):
  - Research Site 5411-0, Bahía Blanca, Buenos Aires
  - Research Site 5414-0, CABA, Buenos Aires
  - Research Site 5405-0, La Plata, Buenos Aires
  - Research Site 5413-0, Mar del Plata, Buenos Aires
  - Research Site 5408-0, Quilmes, Buenos Aires
  - Research Site 5403-0, CABA, Ciudad Autonoma Buenos Aires
  - Research Site 5402-0, Viedma, Río Negro Province
  - Research Site 5401-0, Rosario, Santa Fe Province
  - Research Site 5406-0, Rosario, Santa Fe Province
  - Research Site 5404-0, San Miguel de Tucumán, Tucumán Province
  - Research Site 5407-0, Ciudad Autonoma Buenos Aires
  - Research Site 5409-0, Ciudad Autonoma Buenos Aires
- Australia (13):
  - Research Site 6108-0, Camperdown, New South Wales
  - Research Site 6116-0, Kingswood, New South Wales
  - Research Site 6109-0, Liverpool, New South Wales
  - Research Site 6102-0, Sydney, New South Wales
  - Research Site 6106-0, Birtinya, Queensland
  - Research Site 6101-0, South Brisbane, Queensland
  - Research Site 6107-0, Southport, Queensland
  - Research Site 6104-0, Townsville, Queensland
  - Research Site 6110-0, Adelaide, South Australia
  - Research Site 6103-0, Bendigo, Victoria
  - Research Site 6105-0, St Albans, Victoria
  - Research Site 6113-0, Traralgon, Victoria
  - Research Site 6114-0, Perth, Western Australia
- Belgium (6):
  - Research Site 3201-0, Brussels
  - Research Site 3204-0, Ghent
  - Research Site 3205-0, Jette
  - Research Site 3203-0, Leuven
  - Research Site 3207-0, Liège
  - Research Site 3202-0, Roeselare
- Canada (7):
  - Research Site 1007-0, Winnipeg, Manitoba
  - Research Site 1003-0, Brampton, Ontario
  - Research Site 1001-0, Toronto, Ontario
  - Research Site 1004-0, Montreal, Quebec
  - Research Site 1005-0, Montreal, Quebec
  - Research Site 1006-0, Montreal, Quebec
  - Research Site 1002-0, Sherbrooke, Quebec
- China (55):
  - Research Site 8640-0, Hefei, Anhui
  - Research Site 8614-0, Hefei, Anhui
  - Research Site 8601-0, Beijing, Beijing Municipality
  - Research Site 8625-0, Beijing, Beijing Municipality
  - Research Site 8653-0, Beijing, Beijing Municipality
  - Research Site 8627-0, Chongqing, Chongqing Municipality
  - Research Site 8651-0, Fuzhou, Fujian
  - Research Site 8638-0, Xiamen, Fujian
  - Research Site 8630-0, Lanzhou, Gansu
  - Research Site 8604-0, Guangzhou, Guangdong
  - Research Site 8628-0, Guangzhou, Guangdong
  - Research Site 8621-0, Huizhou, Guangdong
  - Research Site 8622-0, Zhuhai, Guangdong
  - Research Site 8615-0, Nanning, Guangxi
  - Research Site, Baoding, Hebei
  - Research Site 8629-0, Baoding, Hebei
  - Research Site 8645-0, Shijiazhuang, Hebei
  - Research Site 8619-0, Harbin, Heilongjiang
  - Research Site 8649-0, Anyang, Henan
  - Research Site 8609-0, Luoyang, Henan
  - Research Site 8648-0, Weihui, Henan
  - Research Site 8605-0, Zhengzhou, Henan
  - Research Site 8623-0, Zhengzhou, Henan
  - Research Site 8637-0, Wuhan, Hubei
  - Research Site 8608-0, Wuhan, Hubei
  - Research Site 8633-0, Xiangyang, Hubei
  - Research Site 8635-0, Changsha, Hunan
  - Research Site 8654-0, Yongzhou, Hunan
  - Research Site 8646-0, Huai'an, Jiangsu
  - Research Site 8607-0, Nanjing, Jiangsu
  - Research Site 8624-0, Xuzhou, Jiangsu
  - Research Site 8631-0, Nanchang, Jiangxi
  - Research Site 8612-0, Changchun, Jilin
  - Research Site 8618-0, Changchun, Jilin
  - Research Site 8644-0, Changchun, Jilin
  - Research Site 8636-0, Dalian, Liaoning
  - Research Site-8636-0, Dalian, Liaoning
  - Research Site 8643-0, Shenyang, Liaoning
  - Research Site 8642-0, Shenyang, Liaoning
  - Research Site 8634-0, Jinan, Shandong
  - Research Site 8613-0, Jining, Shandong
  - Research Site 8610-0, Linyi, Shandong
  - Research Site 8650-0, Weihai, Shandong
  - Research Site 8603-0, Shanghai, Shanghai Municipality
  - Research Site 8602-0, Shanghai, Shanghai Municipality
  - Research Site 8611-0, Xi’an, Shanxi
  - Research Site 8606-0, Chengdu, Sichuan
  - Research Site 8626-0, Neijiang, Sichuan
  - Research Site 8647-0, Zigong, Sichuan
  - Research Site 8617-0, Tianjin, Tianjin Municipality
  - Research Site 8616-0, Ürümqi, Xinjiang
  - Research Site 8632-0, Kunming, Yunnan
  - Research Site 8652-0, Hangzhou, Zhejiang
  - Research Site 8620-0, Hangzhou, Zhejiang
  - Research Site 8641-0, Hangzhou, Zhejiang
- France (17):
  - Research Site 3311-0, Marseille, Bouches-du-Rhône
  - Research Site 3303-0, La Rochelle, Charente Maritime
  - Research Site 3312-0, Besançon, Doubs
  - Research Site 3308-0, Nîmes, Gard
  - Research Site 3314-0, Bordeaux, Gironde
  - Research Site 3305-0, Toulouse, Haute Garonne
  - Research Site 3309-0, Limoges, Haute Vienne
  - Research Site 3304-0, Montpellier, Herault
  - Research Site 3310-0, Saint-Herblain, Loire Atlantique
  - Research Site 3301-0, Angers, Maine Et Loire
  - Research Site 3315-0, Lille, Nord
  - Research Site 3306-0, Bayonne, Pyrenees Atlantiques
  - Research Site 3318-0, Pierre-Bénite, Rhone
  - Research Site 3313-0, Rouen, Seine Maritime
  - Research Site 3307-0, Avignon, Vaculuse
  - Research Site 3302-0, Créteil, Val De Marne
  - Research Site 3316-0, Paris
- Germany (7):
  - Research Site 4907-0, Erlangen, Bavaria
  - Research Site 4909-0, Wiesbaden, Hesse
  - Research Site 4904-0, Bottrop, North Rhine-Westphalia
  - Research Site 4901-0, Witten, North Rhine-Westphalia
  - Research Site 4903-0, Dresden, Saxony
  - Research Site 4905-0, Berlin
  - Research Site 4906-0, Berlin
- Hong Kong (5):
  - Research Site 8504-0, Hong Kong
  - Research Site 8501-0, Hong Kong
  - Research Site 8503-0, Hong Kong
  - Research Site 8502-0, Hong Kong
  - Research Site 8505-0, Hong Kong
- Hungary (6):
  - Research Site 3603-0, Budapest
  - Research Site 3606-0, Győr
  - Research Site 3604-0, Kecskemét
  - Research Site 3602-0, Salgótarján
  - Research Site 3607-0, Tatabánya
  - Research Site 3605-0, Zalaegerszeg
- Israel (10):
  - Research Site 9710-0, Ashdod
  - Research Site 9706-0, Haifa
  - Research Site 9708-0, Haifa
  - Research Site 9702-0, Jerusalem
  - Research Site 9707-0, Jerusalem
  - Research Site 9703-0, Kfar Saba
  - Research Site 9704-0, Petah Tikva
  - Research Site 9709-0, Ramat Gan
  - Research Site 9705-0, Rehovot
  - Research Site 9701-0, Tel Aviv
- Italy (10):
  - Research Site 3908-0, Bergamo
  - Research Site 3907-0, Brescia
  - Research Site 3901-0, Catania
  - Research Site 3903-0, Catanzaro
  - Research Site 3906-0, Milan
  - Research Site 3911-0, Milan
  - Research Site 3904-0, Milan
  - Research Site 3909-0, Napoli
  - Research Site 3902-0, Pavia
  - Research Site 3905-0, Verona
- Poland (7):
  - Research Site 4804-0, Krakow
  - Research Site 4803-0, Lodz
  - Research Site 4801-0, Poznan
  - Research Site 4802-0, Rzeszów
  - Research Site 4807-0, Torun
  - Research Site 4805-0, Warsaw
  - Research Site 4809-0, Wroclaw
- South Korea (14):
  - Research Site 8211-0, Wŏnju, Gangwon-do
  - Research Site 8204-0, Seongnam-si, Gyeonggi-do
  - Research Site 8201-0, Seoul, Gyeonggi-do
  - Research Site 8202-0, Suwon, Gyeonggi-do
  - Research Site 8208-0, Busan
  - Research Site 8212-0, Cheonan
  - Research Site 8209-0, Incheon
  - Research Site 8207-0, Seoul
  - Research Site 8213-0, Seoul
  - Research Site 8206-0, Seoul
  - Research Site 8210-0, Seoul
  - Research Site 8203-0, Seoul
  - Research Site 8205-0, Seoul
  - Research Site 8214-0, Ulsan
- Spain (18):
  - Research Site 3403-0, Sant Cugat del Vallès, Barcelona
  - Research Site 3409-0, Santiago de Compostela, La Coruña
  - Research Site 3406-0, Majadahonda, Madrid
  - Research Site 3411-0, Pozuelo de Alarcón, Madrid
  - Research Site 3405-0, Pamplona, Navarre
  - Research Site 3410-0, Barcelona
  - Research Site 3402-0, Barcelona
  - Research Site 3404-0, Barcelona
  - Research Site 3416-0, Madrid
  - Research Site 3407-0, Madrid
  - Research Site 3414-0, Madrid
  - Research Site 3401-0, Madrid
  - Research Site 3415-0, Málaga
  - Research Site 3418-0, Málaga
  - Research Site 3408-0, Seville
  - Research Site 3413-0, Seville
  - Research Site 3417-0, Seville
  - Research Site 3412-0, Valencia
- Turkey (Türkiye) (9):
  - Research Site 9001-0, Adana
  - Research Site 9002-0, Ankara
  - Research Site 9006-0, Ankara
  - Research Site 9003-0, Ankara
  - Research Site 9004-0, Ankara
  - Research Site 9009-0, Diyarbakır
  - Research Site 9008-0, Istanbul
  - Research Site 9010-0, Izmir
  - Research Site 9007-0, Samsun
- United Kingdom (15):
  - Research Site 4404-0, Truro, Cornwall
  - Research Site 4408-0, London, Greater London
  - Research Site 4411-0, London, Greater London
  - Research Site 4406-0, London, Greater London
  - Research Site 4416-0, London, Greater London
  - Research Site 4409-0, London, Greater London
  - Research Site 4402-0, Manchester, Greater Manchester
  - Research Site 4415-0, Maidstone, Kent
  - Research Site 4414-0, Bath, Somerset
  - Research Site 4410-0, Cardiff, South Glamorgan
  - Research Site 4405-0, Glasgow, Strathclyde
  - Research Site 4416-A, Sutton, Surrey
  - Research Site 4407-0, Leeds, West Yorkshire
  - Research Site 4403-0, Middlesex
  - Research Site 4401-0, Nottingham

IPD SHARING:
Plan to Share IPD: No